CLINICAL TRIAL: NCT01342432
Title: Comparison of Balance Reeducation Plus General Exercises Versus General Exercises Only: Impact on Pain, Function and Postural Control of Low Back Pain Patients
Brief Title: Impact of a Balance Reeducation Protocol on Pain, Function and Postural Control of Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitari Fieo (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Thais Weber Alencar Bojadsen, PhD, Centro Universitário Fieo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008/069241
Record Dates: First submitted 2011-04-04; First posted 2011-04-27 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2009-12

CONDITIONS: Low Back Pain
Keywords: low back pain; balance reeducation; pain; function
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Balance reeducation plus exercise (Experimental): exercises that challenge postural control are performed in addition to general exercises for stretch and strength of abdominal and paraspinal muscles
  Interventions: Other: Balance reeducation plus general exercise
- General exercise only (Other): general exercise for stretch and strength of paraspinal and abdominal muscles
  Interventions: Other: General exercise only

INTERVENTIONS:
Other: General exercise only — exercises for stretch and strength of paraspinal and abdominal muscles
  Other Names: control group
  Arms: General exercise only
Other: Balance reeducation plus general exercise — patients perform balance reeducation exercises in addition to general exercises for stretch and strength of back and abdominal muscles
  Other Names: balance group, intervention group
  Arms: Balance reeducation plus exercise

SUMMARY:
The purpose of this study is to compare the effects of a balance reeducation protocol and an evidenced based protocol on pain, function and postural control of low back pain patients.

DETAILED DESCRIPTION:
Both groups will perform general exercises for back pain (stretch and strength of paraspinal and abdominal muscles, plus exercises to enhance lumbar and pelvic flexibility but the balance or experimental group will perform in addition five minutes of exercises that challenge postural stability in the sitting position. The evolution of the two groups concerning pain level, function and postural control will be compared.

ELIGIBILITY:
Inclusion Criteria:

* must have low back pain longer than three months and age between 40 and 69 years old

Exclusion Criteria:

* balance or neuromuscular disorders, spine surgery, diabetes.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Perceived pain | 5 weeks
  Pain was measured by an Analogic Visual Scale

SECONDARY OUTCOMES:
Function | 5 weeks
  Function was measured by the Roland-Morris Questionnaire
Postural Control | 5 weeks
  Postural control was measured by Functional Reach Test and by posturography

CONTACTS AND LOCATIONS:
Overall Officials: Thais Bojadsen, PhD, Principal Investigator — Centro Universitario Fieo
Locations (1):
- Centro Universitário Fieo, Osasco, São Paulo, Brazil